CLINICAL TRIAL: NCT02523820
Title: Nebulized Corticosteroid for Post Extubation Stridor in Children: A Randomized Double Blind Controlled Trial
Brief Title: Nebulized Corticosteroid for Post Extubation Stridor in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Nattachai Anantasit, Assistant Professor, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ID10-57-18
Record Dates: First submitted 2015-08-06; First posted 2015-08-14 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Stridor
MeSH Terms: conditions — Respiratory Sounds | interventions — Fluticasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fluticasone propionate (Experimental): Fluticasone 1 mg + Normal saline (NSS) upto 4 ml nebulized after extubation
  Interventions: Drug: fluticasone propionate
- placebo (Placebo Comparator): Normal saline (NSS) 4 ml nebulized after extubation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fluticasone propionate — Flixotide 1 mg + NSS upto 4 ml nebulized after extubation. Record vital signs and modified Westley score at 0, 15, 30, 60 min and 2,4,6 hours
  Other Names: Flixotide
  Arms: fluticasone propionate
Drug: Placebo — NSS 4 ml nebulized after extubation. Record vital signs and modified Westley score at 0, 15, 30, 60 min and 2,4,6 hours
  Other Names: normal saline
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and adverse effect of nebulized corticosteroid to prevent post-extubation stridor in children.

DETAILED DESCRIPTION:
The guideline for prevention and treatment of post-extubation stridor in children is inconclusive include Nebulized epinephrine and intravenous corticosteroid. Nebulized corticosteroid is alternative treatment for viral croup. the rationale of this study to evaluate the efficacy of nebulized fluticasone propionate to prevent pediatric post-extubation stridor

ELIGIBILITY:
Inclusion Criteria:

* Children age between 1 month old - 18 year old who was intubated

Exclusion Criteria:

* Palliative care
* Anatomical abnormalities of airway; subglottic stenosis
* Neuromuscular disease with negative inspiratory force < - 30 mmHg
* Need positive pressure after extubation

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
post-extubation stridor | 6 hours
  patient who developed stridor after extubation within 6 hours

SECONDARY OUTCOMES:
treatment failure | 24 hour
  patient who required escalating of respiratory support such as noninvasive positive pressure ventilation or reintubation within 24 hours
adverse events | 24 hour
  hyperglycemia, oral thrust or GI bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Nattachai Anantasit, Assist Prof., Principal Investigator — Ramathibodi Hospital, Mahidol University
Locations (1):
- Department of Pediatric,Ramathibodi Hospital, Bangkok, Thailand

REFERENCES:
- [Result] Prasertsan P, Nakju D, Lertbunrian R, Chantra M, Anantasit N. Nebulized Fluticasone for Preventing Postextubation Stridor in Intubated Children: A Randomized, Double-Blind Placebo-Controlled Trial. Pediatr Crit Care Med. 2017 May;18(5):e201-e206. doi: 10.1097/PCC.0000000000001124. PMID 28272175